CLINICAL TRIAL: NCT03165721
Title: A Phase II Trial of the DNA Methyl Transferase Inhibitor, SGI-110 (Guadecitabine), In Children And Adults With Wild Type GIST, Pheochromocytoma And Paraganglioma Associated With Succinate Dehydrogenase Deficiency And HLRCC-Associated Kidney Cancer
Brief Title: A Phase II Trial of the DNA Methyl Transferase Inhibitor, Guadecitabine (SGI-110), in Children and Adults With Wild Type GIST,Pheochromocytoma and Paraganglioma Associated With Succinate Dehydrogenase Deficiency and HLRCC-associated Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed to enrollment due to low accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John Glod, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170088; 17-C-0088
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Paraganglioma; Gastrointestinal Stromal Tumors; Carcinoma, Renal Cell; Renal Neoplasms; Pheochromocytoma
Keywords: Renal Cancer; DNA Hypermethylation; Gastrointestinal Stromal Tumors; DNA Methyltransferase (DNMT) Inhibitor; Succinate Dehydrogenase (SDH) Deficiency
MeSH Terms: conditions — Paraganglioma; Gastrointestinal Stromal Tumors; Carcinoma, Renal Cell; Kidney Neoplasms; Pheochromocytoma | interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Patients ≥ 12 Years of Age w/Wild-Type GIST (Experimental): SGI-110 administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle
  Gastrointestinal stromal tumor (GIST)
  Interventions: Drug: SGI-110 (guadecitabine)
- Patients ≥ 12 Years of Age w/PHEO/PGL with SDH-deficient PHE (Experimental): SGI-110 administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle
  Pheochromocytoma and Paraganglioma (PHEO/PGL) with succinate dehydrogenase (SDH)-deficient PHE
  Interventions: Drug: SGI-110 (guadecitabine)
- Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca (Experimental): SGI-110 administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle
  Hereditary leiomyomatosis and renal cell carcinoma (HLRCC)-associated Renal Cell Ca
  Interventions: Drug: SGI-110 (guadecitabine)

INTERVENTIONS:
Drug: SGI-110 (guadecitabine) — SGI-110 will be administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle. Cycles may be repeated until there is evidence of tumor progression clinically or by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or there is intolerable toxicity that is not alleviated by dose reduction.
  Other Names: guadecitabine

SUMMARY:
Background:

Wild-type gastrointestinal stromal tumor (GIST) is a cancer in the esophagus, stomach, or intestines. It does not respond well to standard chemotherapy or radiation therapy. Most people with GIST are treated with imatinib. But it may not work in many children with GIST. Researchers think the drug SGI-110 may help treat people with GIST, pheochromocytoma and paraganglioma (PHEO/PGL), or kidney cancer related to hereditary leiomyomatosis and renal cell carcinoma (HLRCC).

Objective:

To learn if SGI-110 causes GIST tumors to shrink or slows their growth. Also to test how it acts in the body.

Eligibility:

People ages 12 and older who have GIST, PHEO/PGL, or HLRCC that has not responded to other treatments

Design:

Participants will be screened with:

* Physical exam
* Urine tests
* Computed tomography (CT) or magnetic resonance imaging (MRI), or fluorodeoxyglucose (FDG)-positron emission tomography (PET) scan: A machine takes pictures of the body.
* Blood tests

Participants will be injected with SGI-110 under the skin each day for 5 days. This cycle will repeat every 28 days. The cycles repeat until their side effects get too bad or their cancer gets worse.

Participants will have tests throughout study:

* Physical exam and blood and urine tests before each cycle
* Blood tests on days 1, 7, 14, and 28 of the first cycle.
* Scans before cycle 1 and then every other cycle.
* Questionnaires about their pain and quality of life
* Tumor biopsy for those 18 and older: A needle removes a small piece of tumor.

After they stop treatment, participants will have a final visit. This includes an evaluation of their health, pain, and quality of life.

...

DETAILED DESCRIPTION:
Background

* Loss of activity of the Krebs cycle components succinate dehydrogenase (SDH) complex or fumarate hydratase (FH), has been identified as a mechanism of tumorigenesis in subsets of gastrointestinal stromal tumor (GIST), pheochromocytoma and paraganglioma (PHEO/PGL), and renal cell carcinoma.
* Deoxyribonucleic acid (DNA) hypermethylation has been demonstrated in these cancers. Loss of activity of SDH or FH leads to accumulation of the metabolites succinate and fumarate, respectively. Succinate and fumarate act as inhibitors of a broad array of alpha-ketoglutarate dependent dioxygenases. The Ten-eleven Translocation (TET) family of alphaKG-dependent dioxygenase enzymes convert 5-methylcytosine to 5-hydroxymethylcytosine leading to DNA demethylation. Inhibition of these enzymes due to SDH and FH deficiency causes DNA hypermethylation and has been verified in preclinical models.
* Gastrointestinal stromal tumors (GISTs) are the most common mesenchymal tumor of the gastrointestinal tract, resistant to cytotoxic chemotherapy and radiation therapy. KIT and Platelet Derived Growth Factor Receptor Alpha (PDGFRA) mutations have been identified as tumor initiating events in 85% of adult patients with GIST and these tumors are responsive to the tyrosine kinase inhibitor, Imatinib. In pediatric patients, however, 85% of GISTs lack KIT and PDGFRA mutations (wild-type) and imatinib is not effective.
* Recent work in the Pediatric and Wild-Type (wt) GIST Clinic at the National Cancer Institute (NCI) led to the identification of succinate dehydrogenase (SDH) deficiency in approximately 90% of wildtype GIST.
* In addition to wild-type GIST, SDH deficiency is also present in 30% of pheochromocytoma and paraganglioma (PHEO/PGL) and a subset of renal carcinoma. Loss of succinate dehydrogenase complex iron sulfur subunit B (SDHB) protein expression is seen in PHEO/PGL and wtGIST either due to mutation in SDH subunit genes or hypermethylation of the SDHC promoter region.
* Mutations leading to loss of function of FH have been identified in PHEO/PGL as well as type II papillary renal cell carcinoma in patients with hereditary leiomyomatosis and renal cell cancer (HLRCC). An FH-deficient paraganglioma had DNA hypermethylation as demonstrated by array and immunohistochemistry showed increased 5hmC levels in paragangliomas and pheochromocytomas.
* SGI-110 is a small molecule derivative of decitabine that acts as a DNA methyltransferase (DNMT) inhibitor and is resistant to inactivation by cytidine deaminase, hence may thus have a more favorable pharmacokinetic profile compared to decitabine. Subcutaneously administered SGI-110 is gradually converted to decitabine resulting in prolonged exposure with a several fold increase in apparent T1/2 compared to intravenous decitabine. SGI-110 has been demonstrated in preclinical models to induce a dose-dependent decrease in global DNA methylation and up-regulate expression of specific genes including Melanoma-associated antigen 1 (MAGE-A1) and New York esophageal squamous cell carcinoma 1 (NY-ESO-1) through decreased methylation.
* We are proposing a phase II trial with SGI-110 in these SDH-deficient and fumarate hydratase (FH)-deficient tumors.

Objectives:

-To assess the clinical activity of SGI-110 in patients with wt-GIST, SDH-deficient PHEO/PGL, and HLRCC-associated renal cell carcinoma (RCC) using Response Evaluation Criteria in Solid Tumors (RECIST).

Eligibility:

* Adults and children (greater than or equal to 12 years of age) with wt-type GIST, SDH deficient PHEO/PGL, or HLRCC-associated RCC and measurable disease will be eligible.
* Newly diagnosed patients with PHEO/PGL or HLRCC-associated RCC with localized, resectable disease will not be eligible. Patients with PHEO/PGL or HLRCC-associated RCC with unresectable localized disease and/or metastatic disease will be eligible.
* Newly diagnosed patients with wt-GIST with completely resectable disease will not be eligible. Patients with wt-GIST with metastatic disease and/or residual or recurrent tumor following surgical debulking will be eligible
* Patients with wt-GIST or HLRCC-associated RCC who have not previously received systemic therapy are eligible as there are no standard chemotherapy regimens known to be effective for these cancers.
* Must have adequate performance status, may not be pregnant or breastfeeding, and must have adequate major organ function.
* No history of severe or uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic cardiovascular or pulmonary disease will be excluded.

Design:

* This is a single site, open label, phase II study using a small optimal two-stage design to evaluate the clinical response in three groups of patients:

  1. wild-type GIST (GIST without KIT or PDGFRA mutation)
  2. PHEO/PGL in patients with germline SDH subunit mutation, or
  3. RCC associated with HLRCC
* SGI-110 will be administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle to the three groups of patients.
* SGI-110 activity will be assessed by imaging response of measurable disease using Response Evaluation Criteria in Solid Tumors (RECIST)v1.1, using computed tomography (CT), magnetic resonance imaging (MRI) and/or positron emission tomography (PET).
* Patients will be closely monitored for development of toxicity with regular physical examinations and laboratory evaluations. Toxicity will be graded using version 4.0 of the National Cancer Institute (NCI) Common Toxicity Criteria.
* SGI-110 related toxicities greater than or equal to grade 3 will be considered treatment limiting toxicities, unless they are reversible within 72 hours with supportive care. Following recovery from toxicity up to 2 dose reductions will be allowed.
* Initially 7 evaluable patients in each group (strata) will be enrolled and if 0 of the 7 have a response, then no further patients will be accrued in that strata. If 1 or more the first 7 (14.3% or more) have a response, then accrual would continue until a total of 21 patients have enrolled in that strata. If at least 3 responses (at least 14.3%) are observed among the 21 evaluable patients, the agent should be considered worthy of further testing in this disease.
* Enrolling 2 patients/month, it is estimated to require 3 years to complete accrual to a maximum of 70 patients, a maximum of 63 evaluable patients allowing for a small number (7) of inevaluable patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must:

* Have recurrent or refractory/unresectable disease for which there is no known curative therapy.

  ---Wild type-gastrointestinal stromal tumors (GIST): Patients with recurrent or progressive disease will be eligible. Newly diagnosed patients with resectable localized disease will not be eligible. Newly diagnosed patients with metastatic disease and newly diagnosed patients with residual tumor following surgical debulking will be eligible.
  * Paraganglioma-Pheochromocytoma (PHEO/PGL): Patients with recurrent or progressive disease will be eligible. Newly diagnosed patients with PHEO/PGL that is metastatic at diagnosis and/or unresectable will be eligible Patients with PHEO/PGL with localized (non-metastatic), resectable disease will not be eligible.
  * Renal cell cancer associated with HLRCC: Patients with localized, resectable HLRCC-associated renal cell cancer will not be eligible. Patients with metastatic and/or unresectable Hereditary leiomyomatosis and renal cell cancer (HLRCC)-associated renal cell cancer will be eligible.
* Have one of the following confirmed histologically, cytologically, or through biochemical testing:

  * wild-type GIST (GIST without KIT or platelet derived growth factor receptor alpha (PDGFRA) mutation);
  * PHEO/PGL with a germline mutation in Succinate Dehydrogenase Complex Flavoprotein Subunit A (SDHA), Succinate Dehydrogenase Complex Flavoprotein Subunit B (SDHB), SDHC, or SDHD;

    --renal cell cancer associated with HLRCC.
* Testing will be performed in Clinical Laboratory Improvement Amendments (CLIA) certified labs using genetic tests for KIT/PDGFRA and testing panels developed for patients with PHEO/PGL. Results from outside labs will be accepted. Pathologic diagnosis will be reviewed and verified at the Clinical Center.
* Age: be greater than or equal to 12 years of age

Because there is no dosing or adverse event data currently available on the use of SGI-110 in children < 18 year of age, children < 12 years of age will be excluded from this study, but may be eligible for future pediatric trials should the results of the study be positive.

- Measurable disease:

Have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as greater than or equal to 20 mm with conventional techniques or as greater than 10 mm with spiral computed tomography (CT) scan.

* Prior Therapy
* Prior therapy requirements:

  ---Wt-GIST: Because there are no standard chemotherapy regimens known to be effective for wt-GIST, previously untreated participants are eligible.

  --PHEO/PGL with germline SDH subunit mutation: 131I-MIBG in patients with MIBG avid tumors or cytotoxic chemotherapy (cyclophosphamide, vincristine, and dacarbazine (CVD) or temozolomide) is required prior to enrollment on this trial. However, patients who have refused cytotoxic chemotherapy or for whom treatment on this protocol prior to receiving cytotoxic chemotherapy is felt to be in the best interest for the patient by the local investigator will also be eligible.

  ---HLRCC-associated renal cell cancer: Because there are no standard chemotherapy regimens known to be effective for HLRCC-associated renal cell cancer, previously untreated participants are eligible.
* Prior therapy wash-out period requirements

  --Participants must be at least 4 weeks from prior surgical procedures and surgical incisions must be healed.

  ---Participants must have had their last fraction of external beam radiation therapy at least 4 weeks prior to enrollment. Participants with prior radiation therapy must be at least 4 weeks post therapy and have had progression of disease outside the radiation port.
  * Participants must have had their last dose of cytotoxic chemotherapy at least 28 days prior to enrollment, their last dose of biological therapy, such as biological response modifiers (e.g., cytokines), immunomodulatory agents, vaccines, differentiating agents, used to treat their cancer at least 28 days prior to enrollment, their last dose of a monoclonal antibody at least 28 days prior to enrollment, and their last dose of any investigational agent at least 28 days prior to enrollment.
  * Participants must have recovered from the acute toxic effects of prior therapy to a grade 1 level prior to enrollment (does not apply to alopecia).
* Performance Level: Eastern Cooperative Oncology Group (ECOG) performance status less than or equal 2 or Karnofsky greater than or equal to 60% in patients greater than 16 years of age, Lansky greater than or equal to 60 for patients less than or equal to 16 years of age.
* Have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin within normal institutional limits
  * Aspartate aminotransferase (AST) Serum glutamic oxaloacetic transaminase(SGOT)/Alanine aminotransferase (ALT) Serum glutamic pyruvic transaminase(SGPT) less than or equal to 2.5 x institutional upper limit of normal
  * creatinine within normal institutional limits

OR

----creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.

-Birth Control:

The effects of SGI-110 on the developing human fetus are unknown. For this reason and because decitabine is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for 6 months following participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

-Ability of subject or legal guardians (if the patient is <18 years old) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Patients with any one the following will be excluded:

* Ongoing radiation therapy, chemotherapy, hormonal therapy directed at the tumor, immunotherapy, or biologic therapy, including investigational agents for their disease.
* History of allergic reactions to SGI-110 or decitabine.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, symptomatic pulmonary disease or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding

Pregnant women are excluded from this study because SGI-110 is a derivative of decitabine which has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SGI-110, breastfeeding should be discontinued if the mother is treated with SGI-110.

These potential risks may also apply to other agents used in this study.

* Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses, or renal transplant, including any patient known to have hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) will be excluded. Patients with HIV who have adequate cluster of differentiation 4 (CD4) count, not requiring antiretroviral medication, may be enrolled.
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Glod, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ligon JA, Sundby RT, Wedekind MF, Arnaldez FI, Del Rivero J, Wiener L, Srinivasan R, Spencer M, Carbonell A, Lei H, Shern J, Steinberg SM, Figg WD, Peer CJ, Zimmerman S, Moraly J, Xu X, Fox S, Chan K, Barbato MI, Andresson T, Taylor N, Pacak K, Killian JK, Dombi E, Linehan WM, Miettinen M, Piekarz R, Helman LJ, Meltzer P, Widemann B, Glod J. A Phase II Trial of Guadecitabine in Children and Adults with SDH-Deficient GIST, Pheochromocytoma, Paraganglioma, and HLRCC-Associated Renal Cell Carcinoma. Clin Cancer Res. 2023 Jan 17;29(2):341-348. doi: 10.1158/1078-0432.CCR-22-2168. PMID 36302175
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0088.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients ≥ 12 Years of Age w/Wild-Type GIST: SGI-110 administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle
  Gastrointestinal stromal tumor (GIST)
  SGI-110 (guadecitabine): SGI-110 will be administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle. Cycles may be repeated until there is evidence of tumor progression clinically or by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or there is intolerable toxicity that is not alleviated by dose reduction.
- Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE: SGI-110 administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle
  Pheochromocytoma and Paraganglioma (PHEO/PGL) with succinate dehydrogenase (SDH)-deficient PHE
  SGI-110 (guadecitabine): SGI-110 will be administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle. Cycles may be repeated until there is evidence of tumor progression clinically or by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or there is intolerable toxicity that is not alleviated by dose reduction.
- Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca: SGI-110 administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle
  Hereditary leiomyomatosis and renal cell carcinoma (HLRCC)-associated Renal Cell Ca
  SGI-110 (guadecitabine): SGI-110 will be administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle. Cycles may be repeated until there is evidence of tumor progression clinically or by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or there is intolerable toxicity that is not alleviated by dose reduction.
Period: Overall Study
Arm/Group | Patients ≥ 12 Years of Age w/Wild-Type GIST | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca
Started | 7 | 1 | 1
Completed | 3 | 1 | 1
Not Completed | 4 | 0 | 0
Not completed — Refused further treatment | 3 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients ≥ 12 Years of Age w/Wild-Type GIST | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca | Total
Number analyzed (Participants) | 7 | 1 | 1 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 1 | 1 | 9
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.86 (16.03) | 41 (0) | 23 (0) | 34.22 (14.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 0 | 6
  Male | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 4 | 1 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 5 | 0 | 1 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 1 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Overall Response (Complete Response or Partial Response) of SGI-11 Using the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Clinical activity of SGI-11 was assessed using the RECISTv1.1. Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: After the first 4 weeks, then every 8 weeks up to 65 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patients ≥ 12 Years of Age w/Wild-Type GIST | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 7 | 1 | 1
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0

2. Secondary Outcome: Change in Distress From Baseline
Description: Change in distress from baseline was assessed by The Distress Thermometer (DT) visual analog scale. An overall score is derived from specific physical, emotional and family issues identified by the participant to be stressful. No distress (0-4), moderate stress (5) and high distress (6-10).
Time Frame: Baseline, end of cycle 4, and post therapy follow up, approximately 30 days after the final dose of study drug
Population: n=6 for the first Group at the end of cycle 4; this time data at this time point was not collected for one participant. Participant off therapy due to progressive disease (PD) at the end of cycle 1 for the third Group.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Patients ≥ 12 Years of Age w/Wild-Type GIST | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 7 | 1 | 1
Scores on a scale
  Baseline | 6.4 (1.4) | 7 | 2
  End of cycle 4: number analyzed (Participants) | 6 | 1 | 0
  End of cycle 4 | 4.5 (1.5) | 2 |
  Post therapy follow up, approximately 30 days after the final dose of study drug: number analyzed (Participants) | 7 | 1 | 0
  Post therapy follow up, approximately 30 days after the final dose of study drug | 4.1 (2.4) | 3 |

3. Post Hoc Outcome: Progression Free Survival Probability at 6 Months
Description: Time interval from start of treatment to documented evidence of disease progression. Progression were evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Disease progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progressions.
Time Frame: 6 months
Population: Patient's progressed at 3.9 months and 1.1 month respectively, for the second and third groups.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Patients ≥ 12 Years of Age w/Wild-Type GIST | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 7 | 1 | 1
Percent probability | 85.7 [33.4 to 97.9] | 0 | 0

4. Post Hoc Outcome: Progression Free Survival (PFS) Probability at 12 Months
Description: as for outcome 3
Time Frame: 12 months
Population: Patient's progressed at 3.9 months and 1.1 month respectively, for the second and third groups.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Patients ≥ 12 Years of Age w/Wild-Type GIST | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 7 | 1 | 1
Percent probability | 53.6 [13.2 to 82.5] | 0 | 0

5. Post Hoc Outcome: Overall Survival (OS)
Description: Time from treatment start date until date of death or date last known alive.
Time Frame: Time from treatment start date until date of death or date last known alive, up to approximately 3 years, 2 months.
Reporting Status: Not Posted, anticipated posting 2026-02

6. Post Hoc Outcome: Quality of Life (QOL) Relative to Any Degree of Response (Patient-Reported Outcomes Measurement Information System (PROMIS) Global Physical Health)
Description: Quality of Life (QOL) was assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Physical Health. Overall scores were derived from five quality of life domains: physical function, pain interference, fatigue, emotional health and social health). T-Score distributions are standardized so that a score of 50 represents the mean for the US general population with a standard deviation around that mean of 10 points.
Time Frame: Baseline, at the end of cycle 4, and post therapy follow up, approximately 30 days after the final dose of study drug
Population: Participant off therapy due to progressive disease (PD) at the end of cycle 1 in the third Group.
Measure: Mean (95% Confidence Interval); unit: t-score
Arm/Group | Patients ≥ 12 Years of Age w/Wild-Type GIST | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 7 | 1 | 1
t-score
  Baseline | 45.9 [40.5 to 51.3] | 54.1 | 57.7
  End of cycle 4 | 46.5 [40.6 to 52.4] | 61.9 | NA [NA to NA] — Participant off therapy due to progressive disease (PD) at the end of cycle 1.
  Post therapy follow up, approximately 30 days after the final dose of study drug | 44.2 [37.5 to 50.9] | 54.1 | NA [NA to NA] — Participant off therapy due to progressive disease (PD) at the end of cycle 1.

7. Post Hoc Outcome: Quality of Life (QOL) Relative to Any Degree of Response (Patient-Reported Outcomes Measurement Information System (PROMIS) Global Mental Health)
Description: Quality of Life (QOL) was assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Mental Health. Overall scores were derived from five quality of life domains: physical function, pain interference, fatigue, emotional health and social health). T-Score distributions are standardized so that a score of 50 represents the mean for the US general population with a standard deviation around that mean of 10 points.
Time Frame: Baseline, at the end of cycle 4, and post therapy follow up, approximately 30 days after the final dose of study drug
Population: n=6 for the first Group at the end of cycle 4; this time data at this time point was not collected for one participant. Participant off treatment at cycle 1 due to progressive disease (PD) in the third Group.
Measure: Mean (95% Confidence Interval); unit: t-score
Arm/Group | Patients ≥ 12 Years of Age w/Wild-Type GIST | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 7 | 1 | 1
t-score
  Baseline | 43.2 [39.7 to 46.7] | 41.1 | 62.5
  End of cycle 4: number analyzed (Participants) | 6 | 1 | 0
  End of cycle 4 | 46.0 [41.9 to 50.1] | 53.3 |
  Post therapy follow up, approximately 30 days after the final dose of study drug: number analyzed (Participants) | 7 | 1 | 0
  Post therapy follow up, approximately 30 days after the final dose of study drug | 41.2 [36.8 to 45.6] | 45.8 |

8. Post Hoc Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approx. 1 mos and 5 days for the Gastrointestinal stromal tumor (GIST) group; 3 mos and 25 days for the Pheochromocytoma/Paraganglioma (Pheo/PGL) group;and 30 mos and 2 days for the Renal Cell Cancer group.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients ≥ 12 Years of Age w/Wild-Type GIST | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 7 | 1 | 1
Participants | 7 | 1 | 1

9. Post Hoc Outcome: Maximum Observed Plasma Concentration (Cmax) of Guadecitabine (SGI-110)
Description: The maximum observed analyte concentration in serum was reported.
Time Frame: Prior to first dose in cycle 1 and at 0.5 hour (+/- 15 minutes), 1 hour (+/- 15 minutes), 2 hour (+/-30 minutes), 4 hour (+/- 30 minutes), 6 hour (+/- 1 hour) and 24 hours (+/- 2 hours) after the first dose of drug in Cycle 1.
Population: Data was analyzed together for all participants because tumor type would not be expected to impact pharmacokinetic parameters or measures of pharmacodynamics that use peripheral blood mononuclear cells (LINE-1 demethylation).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Patients≥12 Years of Age w/Wild-Type GIST, SDH-deficient PHEO/PGL, or HLRCC-associated Renal Cell Ca: Gastrointestinal stromal tumor (GIST); Pheochromocytoma and Paraganglioma (PHEO/PGL) with succinate dehydrogenase (SDH)-deficient PHE; or Hereditary leiomyomatosis and renal cell carcinoma (HLRCC)-associated Renal Cell Ca
  SGI-110 administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle
  SGI-110 (guadecitabine): SGI-110 will be administered subcutaneously at 45mg/m^2/day x 5 days on a 28-day cycle. Cycles may be repeated until there is evidence of tumor progression clinically or by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or there is intolerable toxicity that is not alleviated by dose reduction.
Arm/Group | Patients≥12 Years of Age w/Wild-Type GIST, SDH-deficient PHEO/PGL, or HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 9
ng/mL | 45 (42.7)

10. Post Hoc Outcome: Percent Decrease in Long Interspersed Nuclear Element -1 (LINE-1) Demethylation
Description: Percent decrease from baseline in long interspersed nuclear element -1 (LINE-1) demethylation in peripheral blood mononuclear cells (PBMC) using pyrosequencing and urine and plasma glycolytic metabolites.
Time Frame: Day 14 of cycle 1
Population: Data was analyzed together for all patients because tumor type would not be expected to impact pharmacokinetic parameters or measures of pharmacodynamics that use peripheral blood mononuclear cells (LINE-1 demethylation).
Measure: Mean (90% Confidence Interval); unit: Percent decrease
Arm/Group | Patients≥12 Years of Age w/Wild-Type GIST, SDH-deficient PHEO/PGL, or HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 2
Percent decrease | 45 [42.2 to 47.8]

11. Post Hoc Outcome: Half Life (t1/2) of Guadecitabine (SGI-110)
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Number; unit: hrs
Arm/Group | Patients≥12 Years of Age w/Wild-Type GIST, SDH-deficient PHEO/PGL, or HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 2
hrs
  Patient 2: number analyzed (Participants) | 1
  Patient 2 | 1.73
  Patient 3: number analyzed (Participants) | 1
  Patient 3 | 1.35

12. Post Hoc Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Guadecitabine (SGI-110)
Description: Time it takes Guadecitabine (SGI-110) the reach the maximum concentration in plasma.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Patients≥12 Years of Age w/Wild-Type GIST, SDH-deficient PHEO/PGL, or HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 9
hr | 4.0 [1.0 to 5.5]

13. Post Hoc Outcome: Area Under the Concentration Time Curve (AUC 0-5hr)
Description: The AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Patients≥12 Years of Age w/Wild-Type GIST, SDH-deficient PHEO/PGL, or HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 9
hr*ng/mL | 114.1 (48.1)

14. Post Hoc Outcome: V(2)/F (Apparent Volume of Distribution)
Description: Apparent volume of distribution is the theoretical volume that would be necessary to contain the total amount of an administered drug at the same concentration that it is observed in the blood plasma.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Number; unit: L
Arm/Group | Patients≥12 Years of Age w/Wild-Type GIST, SDH-deficient PHEO/PGL, or HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 2
L
  Patient 2: number analyzed (Participants) | 1
  Patient 2 | 1127
  Patient 3: number analyzed (Participants) | 1
  Patient 3 | 1147

15. Post Hoc Outcome: (CL/F) Apparent Total Body Clearance
Description: Apparent total body clearance is the time it takes for all Guadecitabine (SGI-110) to be removed from the body.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Number; unit: L/hr
Arm/Group | Patients≥12 Years of Age w/Wild-Type GIST, SDH-deficient PHEO/PGL, or HLRCC-associated Renal Cell Ca
Number analyzed (Participants) | 2
L/hr
  Patient 2: number analyzed (Participants) | 1
  Patient 2 | 452
  Patient 3: number analyzed (Participants) | 1
  Patient 3 | 588

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 1 month and 5 days for the Gastrointestinal stromal tumor (GIST) group, 3 months and 25 days for the Pheochromocytoma and Paraganglioma (Pheo/PGL) group, and 30 months and 2 days for the Renal Cell Cancer group.
Arm/Group | Patients ≥ 12 Years of Age w/Wild-Type GIST | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 4/7 | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 7/7 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients ≥ 12 Years of Age w/Wild-Type GIST (N=7) | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE (N=1) | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca (N=1)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, Tumor debulking (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients ≥ 12 Years of Age w/Wild-Type GIST (N=7) | Patients ≥ 12 Years of Age w/PHEO/PGL With SDH-deficient PHE (N=1) | Patients ≥ 12 Years of Age w/HLRCC-associated Renal Cell Ca (N=1)
Anemia (Blood and lymphatic system disorders) | 2 (12) | 0 (0) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (Injury, poisoning and procedural complications) | 6 (13) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (7) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 7 (18) | 1 (5) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 7 (26) | 1 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (8) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (8) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (5) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (4) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (6) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (3) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Flashing lights (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 2 (3) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Feeling warm (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (22) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (7) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Investigations - Other, Sinus arrhythmia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (9) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, R. arm Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Weight gain (Investigations) | 4 (6) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT03165721/Prot_SAP_000.pdf
  • Informed Consent Form: Standard (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT03165721/ICF_003.pdf
  • Informed Consent Form: Assent (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT03165721/ICF_004.pdf